CLINICAL TRIAL: NCT00192868
Title: Drug Elution and DIstal Protection During Percutaneous CoronAry Intervention in sT Elevation Myocardial InfarctiON. Acronym: Dedication
Brief Title: Drug Elution and Distal Protection During Percutaneous Coronary Intervention in ST Elevation Myocardial Infarction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEDICATION
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Coronary Artery Disease
Keywords: primary PCI; distal protection; drug eluting stent; restenosis
MeSH Terms: conditions — Coronary Artery Disease | interventions — Drug-Eluting Stents

INTERVENTIONS:
Procedure: Distal protection and drug eluting stent

SUMMARY:
The purpose of this study is to evaluate the clinical, echocardiographic and angiographic outcome of distal protection in the infarct related coronary artery and implantation of drug eluting versus bare metal stents in patients with ST-elevation myocardial infarctions treated acutely with percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Acute onset typical chest pain of < 12 hours' duration
* ST-elevation of > 4 mm (1mm = 0.1 mV) in contiguous leads of the electrocardiogram
* High grade stenosis or occlusion of a native major coronary artery that can be crossed with a soft or intermediate tip guidewire
* Possibility to perform distal protection of the infarct-related artery

Exclusion Criteria:

* History of previous myocardial infarction
* Use of fibrinolytic agents for the index infarction
* Left main stenosis
* Heavily calcification of abdominal aorta or occlusive iliofemoral disease hampering access to the coronary ostias by the femoral route
* Known renal failure
* Other significant cardiac disease
* Other severe disease with an expected survival < 1 year
* Known allergy against clopidogrel or contrast media that can not be avoided/limited by medication
* Linguistic difficulties needing an interpreter
* Gastrointestinal bleeding within 1 month
* Childbearing potential or pregnancy
* Participation in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2005-05; Primary Completion 2009-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
ST segment resolution | 90 min
Late loss (difference between minimal lumen diameter in stented segment immediately after and at 8 month follow up). | immediately after and at 8 month follow up

SECONDARY OUTCOMES:
Restenosis | 8 months
maximal elevations in blood concentrations of CK-MB enzyme and troponin-T | Post procedure
wall motion index | During hospitalisation: day 3-5
Minimal lumen diameter | 8 months
frequency of binary restenosis (>50% diameter stenosis), diameter stenosis (%) in the stented segment. | 8 months
Occurrence of stent thrombosis and MACE. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Henning Kelbaek, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Cardiac Cath Lab, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Kaltoft A, Kelbaek H, Thuesen L, Lassen JF, Clemmensen P, Klovgaard L, Engstrom T, Botker HE, Saunamaki K, Krusell LR, Jorgensen E, Tilsted HH, Christiansen EH, Ravkilde J, Kober L, Kofoed KF, Terkelsen CJ, Helqvist S. Long-term outcome after drug-eluting versus bare-metal stent implantation in patients with ST-segment elevation myocardial infarction: 3-year follow-up of the randomized DEDICATION (Drug Elution and Distal Protection in Acute Myocardial Infarction) Trial. J Am Coll Cardiol. 2010 Aug 17;56(8):641-5. doi: 10.1016/j.jacc.2010.05.009. PMID 20688033
- [Derived] Kaltoft A, Kelbaek H, Klovgaard L, Terkelsen CJ, Clemmensen P, Helqvist S, Lassen JF, Thuesen L. Increased rate of stent thrombosis and target lesion revascularization after filter protection in primary percutaneous coronary intervention for ST-segment elevation myocardial infarction: 15-month follow-up of the DEDICATION (Drug Elution and Distal Protection in ST Elevation Myocardial Infarction) trial. J Am Coll Cardiol. 2010 Mar 2;55(9):867-71. doi: 10.1016/j.jacc.2009.09.052. PMID 20185036
- [Derived] Kelbaek H, Thuesen L, Helqvist S, Clemmensen P, Klovgaard L, Kaltoft A, Andersen B, Thuesen H, Engstrom T, Botker HE, Saunamaki K, Krusell LR, Jorgensen E, Hansen HH, Christiansen EH, Ravkilde J, Kober L, Kofoed KF, Terkelsen CJ, Lassen JF; DEDICATION Investigators. Drug-eluting versus bare metal stents in patients with st-segment-elevation myocardial infarction: eight-month follow-up in the Drug Elution and Distal Protection in Acute Myocardial Infarction (DEDICATION) trial. Circulation. 2008 Sep 9;118(11):1155-62. doi: 10.1161/CIRCULATIONAHA.107.758698. Epub 2008 Aug 25. PMID 18725489
- [Derived] Kelbaek H, Terkelsen CJ, Helqvist S, Lassen JF, Clemmensen P, Klovgaard L, Kaltoft A, Engstrom T, Botker HE, Saunamaki K, Krusell LR, Jorgensen E, Hansen HH, Christiansen EH, Ravkilde J, Kober L, Kofoed KF, Thuesen L. Randomized comparison of distal protection versus conventional treatment in primary percutaneous coronary intervention: the drug elution and distal protection in ST-elevation myocardial infarction (DEDICATION) trial. J Am Coll Cardiol. 2008 Mar 4;51(9):899-905. doi: 10.1016/j.jacc.2007.10.047. PMID 18308157